CLINICAL TRIAL: NCT02382094
Title: Clinical Trial to Study Quality of Life in Prostate Cancer Patients by Randomizing Anti-androgen Versus Total Androgen Blockage Prior to Curative Intended Radiation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, khairul Majumder, MD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RCT-PC-QLS 2004
Record Dates: First submitted 2015-03-05; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Prostate Cancer
Keywords: curative intention; radiation Therapy; health related quality of life
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm AA(anti-androgen) (Experimental): Bicalutamide 150 mg per os daily + if needed Tamoxifen 10 mg against breast tenderness/gynecomasti.
  Interventions: Drug: Bicalutamide
- Arm TAB (Total androgen blockade) (Other): Bicalutamide 50 mg orally daily + Goserelin 3.6 mg subcutaneously every 28±2 days + if needed Tamoxifen 10 mg against breast tenderness/gynecomasti.
  Interventions: Drug: Bicalutamide

INTERVENTIONS:
Drug: Bicalutamide
  Other Names: Casodex

SUMMARY:
Phase III clinical trial to study quality of life in prostate cancer patients by randomizing anti-androgen versus total androgen blockage prior to curative intended radiation therapy.

DETAILED DESCRIPTION:
Primary objective: To study the difference in quality of life in relation to anti-androgen versus total androgen blockage.

Exploratory parameters: ▪ Time to PSA relapse

* Time to symptom giving metastasis
* Overall survival

Patients with localized /locally advanced prostate cancer were subject to treatment with curative intention. They could be divided into three groups according to the risk of metastasis. Mainly intermediate risk group of patients were included in this study. Patients with low risk could be included if they were subject to neo-adjuvant hormonal therapy. Different risk groups were defined as below:

Low risk group: PSA ≤10 ng/ml Gleason score ≤ 6 Tumour stage ≤ T2b Intermediate risk group: Presence of 1-2 factors of high risk. High risk group: PSA >10 ng/ml Gleason score ≥7 Tumour stage T2c - T3b

ELIGIBILITY:
1. Histopathologically verified prostatic adenocarcinoma.
2. All consecutive patients referred for radiation therapy with combination method i.e. both external beam RT and HDR brachytherapy or other fractionation with curative intention.
3. Patients with intermediate risk group of prostate cancer will mainly be included in this study where radiotherapy with intention to cure is indicated and possible to perform. The intermediate risk group is defined as having 1-2 high risk factors for metastasis. Patients with low risk can only be possible to include if there is an indication of neo-adjuvant hormonal therapy.
4. No signs of distant metastasis.
5. Informed consent.

   -

Exclusion Criteria:

1. Failure to fulfill inclusion criteria.
2. Severe hepatic or renal failure, according to clinical and laboratory examinations, serum creatinine > 225 mmol/l.
3. Concomitant diseases that would influence the planned treatment (e.g. Inflammatory bowel disease, urinary incontinence, severe atherosclerosis, myocardial infarction within last 6 months.
4. Previous diagnosis of other malignant diseases excluding patients who are free from relapse after at least 5 years of diagnosis. Patients with basal cell carcinoma are includable.
5. Inability of the patient to cope with the study rules, due to abuses, mentalstatus or other reasons
6. Participation in other clinical studies at the same time if it considers may hamper the assessment of QoL.

   -

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-06; Primary Completion 2009-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 4 years

SECONDARY OUTCOMES:
PSA relapse | 1year
Time to symptom giving metastasis | 1 year
Overall survival | 1 year

REFERENCES:
- [Derived] Majumder K, Nilsson S, Johansson H, Ullen A, Lennernas B, Bergenmar M, Brandberg Y. Higher sexual interest with androgen receptor inhibitor monotherapy than with castration plus an androgen receptor inhibitor in prostate cancer patients treated with curative radiotherapy, but otherwise small health-related quality of life differences: A randomised prospective 18-month follow-up study. Eur J Cancer. 2016 Sep;65:43-51. doi: 10.1016/j.ejca.2016.06.011. Epub 2016 Jul 25. PMID 27459586